CLINICAL TRIAL: NCT05228652
Title: Questionnaire Study to Assess Long-term Psychosocial and Functional Outcomes in Individuals With Virilising Form of Congenital Adrenal Hyperplasia
Brief Title: Questionnaire Study to Assess the Outcomes of the Management of Congenital Adrenal Hyperplasia Individuals
Acronym: CAH-MaS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Arianna Mariotto, Specialty Registrar Paediatric Urology, Manchester University NHS Foundation Trust
Other Study IDs: B01259; 296826 (Other: IRAS)
Record Dates: First submitted 2022-01-07; First posted 2022-02-08 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Adrenal Hyperplasia, Congenital
Keywords: Congenital Adrenal Hyperplasia; feminising clitoroplasty; outcomes of genital surgery in infancy
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected Individuals: Virilised 46XX CAH individuals aged 16 years or above
  Interventions: Other: Questionnaire
- Parents of affected individuals: Parents of virilised 46XX CAH individuals aged 2 years and over.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Three different questionnaires have been developed. They consist of multiple-choice questions and some open-ended questions.
  Other Names: Q1: CAH Management Assessment Questionnaire - Parent; Q2: CAH Management Assessment Questionnaire - Affected Individuals; Q3: Further Questionnaire for Affected Individuals

SUMMARY:
This is a questionnaire study involving women and young girls affected by Congenital Adrenal Hyperplasia (CAH) and their parents. The aim is to obtain information regarding the outcomes of conservative or surgical management of CAH at the Royal Manchester Children's Hospital (RMCH) in the last 50 years, with specific reference to genital appearance and its impact on patient's social/physical/emotional/sexual outcomes. The study wants also investigate on the individuals and parental perspectives on the proposal to take away the option of early childhood surgery for girls with this condition.

DETAILED DESCRIPTION:
Congenital adrenal hyperplasia (CAH) is a heterogeneous group of autosomal-recessive disorders that results in virilisation of the female child due to intrauterine exposure to androgens at a critical phase of differentiation. Female infants may present with a variable degree of genital virilisation, and depending on it and on parental wishes, genital surgery (also called genitoplasty) is offered in infancy/early childhood. Some patients do not undergo surgery in infancy or early childhood, some of these patients may present at a later stage for consideration of genitoplasty, some may request further genitoplasty.

In current practice, most clitoral procedures involve dorsal neurovascular bundle preservation. However, damage to the clitoral innervation through incision could lead to disruption of neurological pathways, compromising clitoral sensitivity, erotic sensation and pleasure.

There is limited and controversial data measuring qualitative outcomes of sexual function and genital sensitivity following feminizing genitoplasty in childhood and it is very important to assess modern surgical and functional outcomes.

Another controversial topic is the timing of surgery, early infancy versus delayed to adolescence/adulthood, when the patient is able to give her opinion.

Currently there is extensive debate at national and international level about the best timing of such surgery and there are proposals to stop funding for all childhood surgery in the above group of children until they are old enough to make a decision.

It is therefore imperative that this decision is informed by evidence, highlighting the importance and necessity of a study that aims to evaluate psychosocial and functional outcomes.

An objective evaluation of outcome of those patients who have been managed under our care - either conservatively or surgically (early or delayed) - would give us data which will be helpful in assessing whether genitoplasty surgery is felt to be necessary by individuals/families and if so, when is the right time to perform it.

It will also usefull to inform NHS England policy and also our consultation with children and their families thus aiding in the decision-making process.

The main objective of this study is to obtain information on psychosocial and functional outcomes and to assess parental and patients' satisfaction with the current approach where parents are given the option of either conservative or surgical management. CAH affected individuals with virilisation of external genitalia raised as females and treated under the care of the team/co-investigators over the last 50 years at RMCH will be identified from the departmental prospective CAH database. They will ask to fill study-specific questionnaires that have been developed by the study committee to explore the study objectives. The questionnaires are directed to CAH affected individuals aged 16 years and over and the parents of CAH affected girls aged 2 years and over. The research will run over a period of 12 months.

The completed questionnaires will be reviewed by a research team member to ensure that the questionnaire is complete and that participants have fully understood the questions. The analysis of the questionnaires will be done by the research team.

ELIGIBILITY:
Inclusion Criteria:

* Parents of CAH affected 46XX individuals aged 2 years and over who were born with virilised genitalia
* CAH affected 46XX individuals who were born with virilised genitalia, 16 years of age and over.

Exclusion Criteria:

* Female DSD children with virilisation which is not due to CAH
* Non-virilised CAH patients
* CAH patients raised as male
* Parents of individuals excluded as above
* Participants who cannot understand questionnaires in English

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: CAH affected individuals aged 16 years and over and parents/guardians of CAH affected girls aged 2 years are eligible for the study.
  All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation except where the study inclusion and exclusion criteria EXPLICITLY state otherwise.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
To assess Individual's and parental view regarding their management using a specific questionnaire | 2 years
  CAH affected individual's and parental satisfaction with the choice and the outcome of their management over the years.

SECONDARY OUTCOMES:
Impact of the condition on individuals | 2 years
  To assess the impact of CAH upon the affected individual's life using a specific questionnaire
The impact of the individual's condition on parents | 2 years
  To assess the impact of CAH upon the parents of affected individual using a specific questionnaire
The impact of the genital appearance on individuals | 2 years
  To assess the impact of genital appearance upon the CAH affected individual's development using a specific questionnaire
The impact of the genital appearance of the individuals on parents | 2 years
  To assess the impact of genital appearance of the CAH affected individual on parents using a specific questionnaire
Impact of the condition on the family. | 2 years
  Parental views on the effect of CAH condition upon the family using a specific questionnaire
Opinion on early childhood surgery. | 2 years
  Parental perspective towards the NHS England proposal to take away the option of early childhood surgery using a specific questionnaire
Opinion on early childhood surgery. | 2 years
  Individual perspective towards the NHS England proposal to take away the option of early childhood surgery using a specific questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Arianna Mariotto, Principal Investigator — Royal Manchester Children's Hospital Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almasri J, Zaiem F, Rodriguez-Gutierrez R, Tamhane SU, Iqbal AM, Prokop LJ, Speiser PW, Baskin LS, Bancos I, Murad MH. Genital Reconstructive Surgery in Females With Congenital Adrenal Hyperplasia: A Systematic Review and Meta-Analysis. J Clin Endocrinol Metab. 2018 Nov 1;103(11):4089-4096. doi: 10.1210/jc.2018-01863. PMID 30272250
- [Background] Baskin LS, Erol A, Li YW, Liu WH, Kurzrock E, Cunha GR. Anatomical studies of the human clitoris. J Urol. 1999 Sep;162(3 Pt 2):1015-20. doi: 10.1016/S0022-5347(01)68052-2. PMID 10458423
- [Background] Binet A, Lardy H, Geslin D, Francois-Fiquet C, Poli-Merol ML. Should we question early feminizing genitoplasty for patients with congenital adrenal hyperplasia and XX karyotype? J Pediatr Surg. 2016 Mar;51(3):465-8. doi: 10.1016/j.jpedsurg.2015.10.004. Epub 2015 Oct 22. PMID 26607969
- [Background] Fagerholm R, Santtila P, Miettinen PJ, Mattila A, Rintala R, Taskinen S. Sexual function and attitudes toward surgery after feminizing genitoplasty. J Urol. 2011 May;185(5):1900-4. doi: 10.1016/j.juro.2010.12.099. PMID 21439585
- [Background] Frost-Arner L, Aberg M, Jacobsson S. Clitoral sensitivity after surgical correction in women with adrenogenital syndrome: a long term follow-up. Scand J Plast Reconstr Surg Hand Surg. 2003;37(6):356-9. doi: 10.1080/02844310310007863. PMID 15328775
- [Background] Lee PA, Witchel SF. Genital surgery among females with congenital adrenal hyperplasia: changes over the past five decades. J Pediatr Endocrinol Metab. 2002 Nov-Dec;15(9):1473-7. doi: 10.1515/jpem.2002.15.9.1473. PMID 12503853
- [Background] Lesma A, Bocciardi A, Corti S, Chiumello G, Rigatti P, Montorsi F. Sexual function in adult life following Passerini-Glazel feminizing genitoplasty in patients with congenital adrenal hyperplasia. J Urol. 2014 Jan;191(1):206-11. doi: 10.1016/j.juro.2013.07.097. Epub 2013 Aug 6. PMID 23933397
- [Background] O'Connell HE, Sanjeevan KV, Hutson JM. Anatomy of the clitoris. J Urol. 2005 Oct;174(4 Pt 1):1189-95. doi: 10.1097/01.ju.0000173639.38898.cd. PMID 16145367
- [Background] Schnitzer JJ, Donahoe PK. Surgical treatment of congenital adrenal hyperplasia. Endocrinol Metab Clin North Am. 2001 Mar;30(1):137-54. doi: 10.1016/s0889-8529(08)70023-9. PMID 11344932
- [Background] Shalaby M, Chandran H, Elford S, Kirk J, McCarthy L. Recommendations of patients and families of girls with 46XX congenital adrenal hyperplasia in the United Kingdom regarding the timing of surgery. Pediatr Surg Int. 2021 Jan;37(1):137-143. doi: 10.1007/s00383-020-04780-3. Epub 2020 Nov 23. PMID 33230638
- [Background] Speiser PW, White PC. Congenital adrenal hyperplasia. N Engl J Med. 2003 Aug 21;349(8):776-88. doi: 10.1056/NEJMra021561. No abstract available. PMID 12930931